CLINICAL TRIAL: NCT02941159
Title: A Phase I Single Blind, Randomized, Placebo Controlled, Parallel Group Study to Investigate the Safety and Tolerability of SF2000SD in Healthy Male Volunteers
Brief Title: SF2000SD Clinical Trial in Zambia
Acronym: SF2000SD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tropical Diseases Research Centre, Zambia (Other Government)
Collaborators: National Institute for Scientific and Industrial Research (Unknown); University of Zambia (Other); National AIDS/TB/STIs Council of Zambia (Unknown); Copperbelt University of Zambia (Unknown); Dr Ludwick Sondashi Formular Clinic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SF2000SDPh1
Record Dates: First submitted 2016-10-08; First posted 2016-10-21 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Good Health

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SF2000SD (Active Comparator): The test product is a Sondashi Formula Spray dried extract (SF2000SD). It is derived from spray drying with water the Sondashi Formula (SF2000), which is a mixture of mixture of 4 plants. SF2000SD is packaged into capsules of 500mg and six capsules are taken twice, daily for 42 days. This drug has anti-HIV properties but in this study we are just looking at safety issues.
  Interventions: Biological: SF2000SD
- Placebo (Placebo Comparator): The placebo arm is composed of capsule containing 500mg of inactive ingredient (Microcrystalline Cellulose PH102 -240mg; Starch - 10mg; Magnesium Stearate -10mg; and Maltodextrin Unidry 20 - 240mg).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: SF2000SD — This is an intergrase inhibitor
  Arms: SF2000SD
Biological: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of SF2000SD in adult male healthy volunteers

DETAILED DESCRIPTION:
INTRODUCTION: Treatment and management of people suffering from HIV, AIDS and opportunistic infections using conventional therapeutic interventions is beyond the reach of most governments because of the cost of imported medicines. The WHO has approved the strategy and promotion of the use of Traditional Medicine in Health Systems.

The primary health care places traditional medicines high on its list of priorities and emphasizes their easy availability and use. There is however a need for scientific validation of most potential medicinal plants available in many poor countries and research must focus on the safety and efficacy of these traditional medicines to support their widespread usage. This study intends to conduct a phase I clinical trial using the SF2000SD.

History of SF2000 use: The Sondashi Formula 2000, code named "SF2000" is a mixture of 4 plants. Patients suffering from HIV/AIDS have been using this traditional medicine for the management of their illness.

JUSTIFICATION:

A more acceptable dosage form i.e. a spray dried extract (SF2000SD) has been developed based on the SF2000 inventor's traditional preparation the commencement of a phase I clinical safety study involving eligible adult male health individual volunteers is warranted. Information will be collected to scientifically ascertain the safety of SF2000 in these volunteers paving the way for a phase II clinical study to be conducted after phase I.

METHODS:

Study design: The study will be a longitudinal clinical trial of adult healthy male volunteers taking SF2000SD or placebo under directly observed therapy (DOT). The study participants will be randomized to each treatment arm as they are being enrolled into the study. Each treatment arm/group A, B and C will have fifteen (15) study participants, total 45. Apart from the PI the other investigators will be blinded to the participants' treatment arms. The study participants will also be blinded to the treatment arms and their contents.

Study site: The study shall be undertaken at the Tropical Diseases Research Centre, Ndola. Study personnel The following personnel will be available.

1. Project administrator
2. Social scientists
3. Research nurses
4. Lab assistants
5. Clinical Officer
6. Medical doctor
7. Pharmacist
8. Specimen Courier staff

Recruitment: Sensitization and awareness posters, volunteer brochures and flyers, direct mailing and presentations will be given to the targeted community. Volunteers will receive further briefing from the Principal Investigator (PI) or Co-Principal Investigator. The briefing will be followed by an opportunity for questions from the volunteers. Potential study participants will be screened for eligibility to participate in the study. All study participants will receive counseling pertaining to their intent to participate in the study from qualified counselors of the research team. Written informed consent which will be validated by the PI or his designee will be obtained from all participants. Forty five (45) healthy males will be recruited into the study.

Method of assigning study participants to treatment arm/group: The blocked randomization method will be used to allocate the participants to the treatment. Selection of participants to each treatment will be based on the rank of 45 randomly generated numbers of sizes between 0 and 1, generated for each sequential participant. Accordingly, participants in blocks of 3 will be ranked according to the random number.

In each block the participants with the highest rank will be allocated to treatment A, the ones with the second highest will be allocated to treatment B, and the ones with the third highest will be allocated to treatment C. A randomization list with participants Identification (ID) numbers will be generated by the statistician and will be kept by the PI. Treatment packs will bear participant ID numbers. Only the PI will know the treatment allocations.

Drug administration: Participants will start taking the dose orally in their respective treatment arms when recruitment for the study is complete. In order to ensure that the study drug is taken, a Directly Observed Treatment (DOT) approach will be used. The study drug will be administered twice daily between 06.00hrs - 09.00hrs and 17.00hrs - 20.00hrs for six weeks. All administrations will be recorded on the dosing sheet and signed by the person administering the treatment and Co-PI or Medical Doctor.

Data Collection: The participants will be required to report any adverse events immediately. At each visit, the participants will also be interviewed on any adverse events since the previous visit. Furthermore, participants will be required to keep a dairy of adverse events for the duration of the study.

The laboratory tests will mainly be carried out at the Tropical Diseases Research Centre (Ndola), and Ndola Central Hospital (Ndola).

The frequency and data collection points at screening, baseline and weeks 1, 3, 6 and 8.

Screening: Week -2 to -1

* Demographic Data and counselling: Demographic data will be recorded and counselling session on HIV testing will be initiated.
* Informed consent: After an in-depth interview, with one study nurse the participant will be asked to document her consent by signing an informed consent. The signed informed consent must be obtained before any tests or evaluations related to the study are carried out.
* Vital Signs: axillary temperature, blood pressure, respiratory rate and pulse, height and weight will be measured.
* Medical history Physical and Clinical Examination: The medical history of the potential participant and general physical examination will be performed.
* Laboratory Tests: HIV, HBV and HCV testing, malaria microscopy, Urinalysis - dipstix, Blood hemoglobin, full blood count and differential, liver and renal function tests will be performed.
* Discharge: Participant will be discharged and will be asked to report one day after at 06:00 hours for the assessment of the eligibility criteria.

Enrolment and study drug administration visit: Week 0

* Vital signs Vital signs will be measured
* Enrolment The Co-PI or the Medical Doctor will assess the eligibility criteria. Eligible participants should have a Karnofsky score of 100% (Appendix XI) The eligible candidate will receive an ID number and will be sent to the study nurse for medication. Non-eligible potential participant will be referred accordingly.
* Medication Study drug will be administered using DOT strategy
* Adverse event and discharge Any adverse event will be recorded, for the details see appendix Discharge after thirty minutes form the time the drug was administered Follow up period: Week 1 to 6
* Adverse Events Report All adverse events will be recorded. Use appendix IV to check for any adverse effects
* Concomitant Medications Any medications taken by the study including traditional medicine subject will be recorded.
* Vital Signs Vital signs will be measured
* Physical and Clinical Examination A general physical examination and a clinical examination will be performed
* Laboratory tests: HIV, HBV and HCV testing, malaria microscopy, Urinalysis - dipstix, Blood hemoglobin, full blood count and differential, liver and renal function tests will be performed.
* Treatment Study drug will be administered; information on medication will be documented including information on any concomitant medication given for the management of adverse events.
* Unscheduled visits throughout follow up during these visits, the same procedures will be applied. Any laboratory study specific or any other measurements can be performed, according to the physician's clinical judgement.

Data Entry: The data generated will be entered and analyzed by STATA computer software.

Statistical Analysis: Null Hypothesis set p-values The SF2000SD herbal preparation is not safe for human consumption P-value = 0.05.

The adverse events will be classified into three to five categories (Adverse events categories against the three "treatments"). Proportions will be compared using the Chi-square test. If the expected frequencies will be less than 5%, then the Fisher's t test will be used. The students' t test will be used to compare the means. The level of statistical significance will be set at 5%.

The clinical findings will also be classified into three to five categories and an exact chi-square test will be done.

If the null hypothesis (no association between occurrence of adverse events or physical examination findings for exact chi-square test and no difference in the changes for analysis of variance test) in the exact Chi-square test or the analysis of variance test is rejected then multiple comparison tests and stratified analysis will be done to compare the placebo against the other treatments.

Conduct interim analysis at week 3 of study starting from baseline (baseline to be all at the same time for all 45 participants if possible - must be included in randomization).

QUALITY CONTROL: The Investigators will review the consent and screening processes with all study stuff prior to commencement of the study to ensure that a standardized approach is followed during the study. In addition, the Investigators will frequently conduct performance assessments of the study support staff to ensure smooth collection of reliable data and review participants' concerns during the study. In addition the study monitor will visit at initiation, during the conduct of the study and at closure to verify if the study is being conducted in compliance with, Protocol/amendment(s), with Good Clinical Practices, Standard Operating Procedures (SOPs) and applicable regulatory requirements.

PROCEDURES TO HANDLE ADVERSE EVENTS: At admission for each treatment period study participants will be instructed to report any changes in normal health that they experience to the Principal Investigator or Co-Principal Investigator. AEs will also be elicited by indirect questioning at regular intervals, usually at the time of measurement of vital signs, with such questions as "How do you feel today? or "Is anything bothering you?" No study participant shall be permitted any medication during the study except as permitted by the study medical doctor.

All AEs or symptoms will be recorded in the CRF. Any SAE will be reported to the Principal Investigator/Co- Principal Investigator, within 48 hours (0977 655096 or 0966 263271), who in turn will report them to the Ethics Committee and DSMB. On the basis of the occurrence and severity of AEs, coupled with results of any other observations, the Principal Investigator or Co-Principal Investigator, at his discretion and in consultation with the DSMB, may decide to withdraw a study participant or prematurely end the study for reasons of clinical safety. The time of such termination will be recorded and palliative treatment will be instituted as needed.

TRIAL STOPPING RULES: The DSMB has the right to stop the trial based on the following rules:

* The occurrence of any major life threatening adverse event may result in the trial being abandoned immediately at the discretion of the DSMB. The investigators together with the DSMB may agree to stop the study should a certain number of participants experience SAE.
* An occurrence of a SAE directly attributed to SF2000SD.
* If any number of participants have abnormal laboratory results or other AEs over Grade 3 as per the exclusion criteria, then this would warrant for the exceptional meeting of the DSMB to determine whether the trial should be stopped.

REASONS FOR NOT COMPLETING THE STUDY: Participants may not complete the study for medical or non-medical reasons PROJECT MANGEMENT: The project will be managed by four investigators: PI, Co-PI (MD), Biostatistician and Social Scientist.

DATA MONITORING: Data Safety Monitoring Board (DSMB) will be responsible to monitor the progression of the study and analyzing the data generated.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in study, the participant should be;

1. Male aged 18 to 45 years.
2. Available in Ndola during the 10 weeks study duration.
3. Able to provide proof of residence.
4. Able to complete Consent Form
5. In good health as determined by the combination of medical history, physical examination, and clinical judgment and laboratory results following TDRC normal ranges. Urine dipstick for protein and blood should be negative or trace. If either is ≥1+, complete urinalysis will be obtained (UA). If microscopic UA confirms hematuria or proteinuria ≥ 1+, the volunteer is ineligible.
6. Serologically negative for HIV, HBV and HCV infection.

Exclusion Criteria:

Anyone who meets ANY of the following exclusion criteria will NOT qualify for enrolment into the study.

1. Female
2. A history related to TB
3. Any of the following chronic illnesses: diabetes, asthma, hypertension, skin conditions.
4. On herbal medicine and/ or traditional medicines or immune boosting treatments
5. Received an investigational drug or herbal medicine not less than 2 months by the time of administration of the study dose
6. excessive alcohol consumption/alcohol abuse
7. Smokes
8. HIV and/or HBV and/or HCV positive

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-11 (Actual); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of study participants with clinical adverse events such as diarrhea, vomiting, changes in vital signs etc. associated with the test product | 56 days
Proportion of study participants with changes in laboratory liver and renal values after administration of test product. These will include ALT, AST, ALP, Total biluribin, Glucose, Urea and Creatinine | 56 days
Proportion of study participants with changes in blood hematological values after administration of test product. This will involve Full Blood Count (FBC) including differential for white blood cells | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Ray Handema, PhD, Principal Investigator — Tropical Diseases Research Centre
Locations (1):
- Tropical Diseases Resaerch Centre, Ndola, Copperbelt, Zambia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Holliday I. Traditional medicines in modern societies: an exploration of integrationist options through East Asian experience. J Med Philos. 2003 Jun;28(3):373-89. doi: 10.1076/jmep.28.3.373.14587. PMID 12815539
- [Background] Arimori S, Nozaki H, Morita K, Arimori K. Case report: the effect of a Chinese herbal medicine, BG-104 in two HIV positive hemophiliacs. Biotherapy. 1993;7(1):55-7. doi: 10.1007/BF01878154. PMID 7915126
- [Background] Timmermans K. Intellectual property rights and traditional medicine: policy dilemmas at the interface. Soc Sci Med. 2003 Aug;57(4):745-56. doi: 10.1016/s0277-9536(02)00425-2. PMID 12821021
- Available data/document: Study Protocol — http://www.tdrc.org.zm — Data documents can be requested from at info@tdrc.org.zm using the above given website contact page